CLINICAL TRIAL: NCT00967798
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Whether Chronic Treatment of Cystic Fibrosis Subjects With Impaired Glucose Tolerance Using Sitagliptin (Januvia) Prevents the Development of Diabetes
Brief Title: Prevention of Cystic Fibrosis Diabetes
Acronym: Prevent
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Could not achieve target enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arlene Stecenko, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00012724; 1R01FD003527-01 (FDA)
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis; Prediabetes
Keywords: cystic fibrosis; diabetes; inflammation; oxidative stress; redox balance; lung disease
MeSH Terms: conditions — Cystic Fibrosis; Prediabetic State; Diabetes Mellitus; Inflammation; Lung Diseases | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental): CF patients receiving Sitagliptin.
  Intervention: Dose is 100 mg taken orally once a day in the morning with breakfast. Duration is one year or until converted to CF diabetes, whichever comes sooner.
  Interventions: Drug: Sitagliptin
- Sugar pill (Placebo Comparator): CF patients receiving placebo.
  Intervention: Placebo is taken orally once a day in the morning with breakfast. Duration is one year or until converted to CF diabetes, whichever comes sooner.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100 mg of sitagliptin is taken orally each morning with breakfast. Duration is 12 months or conversion to CF diabetes, whichever comes first.
  Other Names: Januvia

SUMMARY:
Acute systemic hyperglycemia causes oxidative stress and a pro-inflammatory response. The pro-inflammatory cytokines induced by hyperglycemia are toxic to islet insulin producing cells, and thus worsen glucose intolerance. Patients with cystic fibrosis (CF) have a high prevalence of CF related diabetes (CFRD) and up to 40% of CF adults develop CFRD. During the prediabetic phase in CF, there is progression from normal glucose homeostasis to high risk prediabetes characterized by episodes of acute hyperglycemia after meals and during respiratory exacerbations. The mild hyperglycemia seen in CF patients with high risk prediabetes following a meal would be expected to induce a degree of systemic inflammation and oxidative stress. These repetitive episodes, if left unchecked, could lead to progression of glucose impairment, worsening severity of oxidative stress and inflammation, and ultimately the development of CFRD, all via hyperglycemia-induced toxicity to beta cells. Furthermore, this process may be accelerated in CF because lung disease and resultant respiratory exacerbations are associated with oxidative stress and inflammation and this will further contribute to beta cell damage.

Sitagliptin is a recently approved agent for type 2 diabetes and markedly enhances insulin secretion in the presence of hyperglycemia and has been shown to be effective in preventing postprandial hyperglycemia. The hypothesis to be tested in this project is that sitagliptin will prevent the development of CFRD in CF subjects with high risk prediabetes by blocking postprandial hyperglycemia. The investigators propose a randomized, double-blind, placebo-controlled, multicenter, 15-month longitudinal study in 118 CF subjects with high risk prediabetes to test this hypothesis. Specifically, the investigators aim to show that chronic treatment with sitagliptin: prevents the conversion to diabetes; results in preservation of beta cell function; reduces systemic measures of oxidative stress and inflammation; and slows the rate of progression of lung disease.

Funding Source - FDA Office of Orphan Products Development

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, multicenter study intending to enroll 118 CF subjects aged 13 years of age or older who have high risk prediabetes. High risk prediabetes was defined during the screening visit by performing an oral glucose tolerance test (OGTT) and finding that the fasting plasma glucose level is between 110-125 mg/dl and/or the 2-hour plasma glucose level is between 140 and 199 mg/dl. Upon enrollment, subjects were randomized to receive either sitagliptin or placebo. Each subject was to be followed for 15 months to determine if sitagliptin prevented the conversion to frank diabetes.

The following was to be done at enrollment and every 6 months: an OGTT with collection of blood at 0, 1/2, and 2 hours for measurement of glucose and insulin in order to determine progression of glucose intolerance; collection of blood at time 0 and 2 hours during the OGTT and measurement of systemic redox status, oxidative stress, and degree of inflammation to determine the degree of basal oxidative stress and inflammation as well as the degree of hyperglycemia-induced oxidative stress and inflammation; collection of exhaled breath condensate in a subset of subjects at selected sites at time 0 and 2 hours during the OGTT and measurement of airway redox status, degree of inflammation, and glucose levels to determine basal respiratory tract redox status and inflammation, the degree of hyperglycemia-induced changes in redox status and inflammation, and correlation between plasma and airway glucose levels; collection of blood to determine safety of the study medication (liver and renal function, complete blood count, electrolyte concentrations); and determination of progression of lung disease as defined by the number of respiratory exacerbations severe enough to require hospitalization and the rate of decline in lung function.

The results of two OGTTs performed at least one week apart was used to determine whether the subject had converted from high risk prediabetes to frank diabetes (primary objective). Conversion to CFRD was defined when both OGTTs were abnormal (abnormal is defined as a fasting plasma glucose level greater than 125 mg/dl and/or a 2 hour glucose level greater than 199 mg/dl). The results of measures of redox balance, oxidant stress and inflammation (secondary objectives) would provide biologic plausibility to our concept on the mechanism of action of sitagliptin in preventing the development of CF diabetes.

Hemoglobin-specific A1c fraction (HbA1c) was to be measured half-way between the 6-monthly visits and a rise of more than 0.5% from the enrollment value would result in two OGTT tests done at least one week apart to determine if diabetes has developed. At these interval study visits, blood was also collected to assess the safety of the study drug and, if the subject was female, to determine if pregnancy had occurred.

In the event that diabetes did develop, the study drug (or placebo) was to be stopped and the subject would have completed the study.

In summary, this was a double-blind, placebo-controlled clinical trial to determine whether sitagliptin prevents the conversion of CF subjects with high-risk prediabetes to frank diabetes. If successful, this would be the first treatment modality available to prevent the development of CFRD, a serious and life shortening complication of CF. Unfortunately, the study sites were unable to achieve enrollment targets and the study was prematurely terminated March 31, 2017 because of low enrollment. For those subjects enrolled in the study, there was no safety concerns. Data are currently being analyzed for the subjects that were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 years of age or older at the time of enrollment
* Diagnosis of cystic fibrosis (CF) confirmed by pilocarpine iontophoresis sweat chloride measurements and/or genotyping
* Clinically stable with no lower respiratory tract exacerbation requiring intravenous antibiotics in the three weeks prior to enrollment
* On a stable clinical treatment regimen for at least three weeks prior to enrollment
* Male or female. If female, is not lactating and has a negative pregnancy test at screening. If female of child bearing potential, willing to practice effective birth control (i.e. a method known to decrease the risk of pregnancy to less than 1%)
* Able to understand and provide informed consent
* Willing and able to comply with the study schedule and testing
* High risk prediabetes as defined by high-risk impaired fasting glucose levels of 110-125 mg/dl and/or a 2-hour plasma glucose level of 140 to 199 mg/dl found on an Oral Glucose Tolerance Test performed at screening 8 weeks or less before enrollment
* Available by telephone
* Has literacy and language skills required to fill out study material

Exclusion Criteria:

* Diagnosed with CF related diabetes
* Chronic heart failure with New York Heart Association (NYHA) class III/IV, ejection fraction less than 25%, or receiving digoxin
* Liver disease as defined by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) three times above the upper limit of normal.
* Serum creatinine greater than 1.3 mg/dl for males and greater than 1.1 mg/dl for females or receiving chronic dialysis
* Taking chronic oral or intravenous glucocorticosteroids during the past month
* On insulin therapy during the past month
* CF lung disease severe enough to require daytime chronic oxygen therapy via nasal cannula during the past month
* Unable to perform pulmonary function testing
* History of any illness or condition that, in the opinion of the sponsor might confound the results of the study or pose an additional risk in administering study drug to the subject
* Post lung or liver transplant
* Listed and awaiting organ transplant
* Current drug or alcohol dependency
* Participating in another clinical drug trial or past participant within 30 days of enrollment
* Pancreatic sufficient
* History of acute pancreatitis as documented by characteristic clinical manifestations and elevation of serum amylase and lipase within the last 2 years.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-05; Primary Completion 2017-03-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A Stecenko, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University and Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2010 and August 2016.
Groups:
- Sitagliptin: Participants randomized to receive Sitagliptin
- Placebo: Participants randomized to receive a placebo
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 17 | 16
Completed | 8 | 13
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Population: All participants are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Conversion to Cystic Fibrosis Related Diabetes
Description: The number of participants with conversion to cystic fibrosis related diabetes was determined.
Time Frame: Month 15
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 17 | 16
Participants | 2 | 1

2. Secondary Outcome: Change in Beta-cell Disposition Index
Description: Preservation of beta-cell function was to be assessed with the disposition index, which is a measurement of beta-cell function adjusted for insensitivity to insulin.
Time Frame: Baseline through Month 15
Population: Samples for the serum assays were destroyed when a freezer broke over a weekend and the samples thawed.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Redox Couples Glutathione/Glutathione Disulfide and Cysteine/Cystine
Description: Cysteine (Cys)/cystine (CySS) and glutathione (GSH)/glutathione disulfide (GSSG) redox couples are biomarkers of oxidative stress.
Time Frame: Baseline through Month 12
Population: Samples for the serum assays were destroyed when a freezer broke over a weekend and the samples thawed.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Inflammatory Cytokines
Description: Hyperglycemia causes release of pro-inflammatory cytokines which can further compromise beta-cell function by increasing insulin resistance and by inducing beta-cell apoptosis. Inflammatory cytokines that have been shown to contribute to destruction of beta-cells include interleukin 1 beta (IL-1b), tumor necrosis factor alpha (TNFa), and interleukin 6 (IL-6).
Time Frame: Baseline through Month 12
Population: Samples for the serum assays were destroyed when a freezer broke over a weekend and the samples thawed.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Percent Predicted FEV1
Description: The decline of lung function was assessed with forced expiratory volume (FEV1), which measures how much air is exhaled during one second of a forced exhale. Change is described as the difference in FEV1 at baseline subtracted from FEV1 at the end of treatment study visit. A protocol change during the study reduced the treatment time from 24 months to 12 months. The end of treatment study visit for participants in the early part of the study occurred at 24 months, while the end of treatment visit was a 12 months for participants enrolling later. Negative values indicate a decline in lung function over the course of the study.
Time Frame: Baseline, end of treatment (Month 12 or Month 24)
Population: The participants included in this analysis are limited to those who have a FEV value for the baseline and end of treatment visits.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 8 | 13
percent predicted | -9.7 (29.4) | -8.5 (14.3)

ADVERSE EVENTS:
Time Frame: For this study, the reporting period for adverse events is from the time the subject signs the informed consent form to 90 days after taking the last dose of the study medication, up to 15 months.
Description: Over 90% of the morbidity in cystic fibrosis (CF) is due to respiratory dysfunction and to readily identify an increase in the frequency of respiratory exacerbations, adverse events will be classified as respiratory or non-respiratory events. Respiratory events are defined as any increase in respiratory symptoms and/or signs (increase sputum production, increase in cough, runny or stuffy nose, a cold, decrease in lung function, and/or change in physical findings of the respiratory system).
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 11/17 | 9/16
Other Adverse Events (participants affected / at risk) | 16/17 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=17) | Placebo (N=16)
Hospitalization due to Respiratory Event (Respiratory, thoracic and mediastinal disorders) | 11 (30) | 9 (27) — Respiratory events are defined as any increase in respiratory symptoms (increase sputum production, increase in cough, runny or stuffy nose, a cold, decrease in lung function, and/or change in physical findings of the respiratory system).
Hospitalization due to erythematous maculopapualr rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lithotripsy with stent placement (Renal and urinary disorders) | 1 (1) | 1 (1)
Hospitalization due to osteochondroplasty of femoral neck due to previous motor vehical accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization due to fever and body aches (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=17) | Placebo (N=16)
Respiratory event (Respiratory, thoracic and mediastinal disorders) | 16 (63) | 16 (109) — Respiratory events are defined as any increase in respiratory symptoms and/or signs (increase sputum production, increase in cough, runny or stuffy nose, a cold, decrease in lung function, and/or change in physical findings of the respiratory system)
Abdominal pain (General disorders) | 2 (2) | 2 (3)
Abnormal lab results (General disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ankle injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0)
Athletes foot (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacterial vaginosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Broken/fractured hand bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Complications with PICC line (Surgical and medical procedures) | 3 (3) | 0 (0)
Complications with port (Surgical and medical procedures) | 1 (2) | 0 (0)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Difficulty sleeping (General disorders) | 1 (2) | 0 (0)
Ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0)
Elevated bilirubin (General disorders) | 1 (1) | 0 (0)
Elevated CO2 (General disorders) | 0 (0) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 1 (1) | 2 (3)
Elevated potassium (Renal and urinary disorders) | 1 (1) | 0 (0)
Elevated eosinophils (General disorders) | 1 (1) | 0 (0)
Elevated lipid panel/triglycerides (General disorders) | 0 (0) | 1 (2)
Elevated prothrombin induced by vitamin K absence-II (PIVKA-II) (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 2 (2) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Head tingling (General disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
hydroceles with scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Increased thirst and urination (General disorders) | 0 (0) | 1 (1)
Intestinal blockage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach blockage with abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness in hands (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kidney stones with colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Migraine headache (General disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neck pain from pulled muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Open wound to left forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostratitis with hematuria (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Right knee contusion with edema (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sebaceous cyst, carbuncle on back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Skin irritation from colistin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sleeplessness, restlessness, bruising, and muscle tightness (General disorders) | 0 (0) | 1 (1)
Tendinitis due to levaquin (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tongue numbness due to colistin (General disorders) | 1 (2) | 0 (0)
Tooth abcess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vomiting and diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight loss (General disorders) | 1 (1) | 3 (3)
Wisdom teeth extraction (Surgical and medical procedures) | 0 (0) | 2 (2)
Yeast infection (Infections and infestations) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Poor enrollment lead to early termination of the study and a small sample size for analyses. Equipment failure resulted in loss of serum samples for some of the secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT00967798/Prot_SAP_000.pdf